CLINICAL TRIAL: NCT00190970
Title: The Effect of Ruboxistaurin Mesylate (LY333531) on Small Fiber Function as Measured by Microvascular Skin Blood Flow, C-Fiber Quantitations in Skin and Quantitative Sensory Testing of Cold and Heat.
Brief Title: The Effect of Ruboxistaurin on Small Fiber Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7550; B7A-MC-MBDO
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — ruboxistaurin

INTERVENTIONS:
Drug: Ruboxistaurin

SUMMARY:
To determine the effect of Ruboxistaurin on small fiber function.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Type 1 or Type 2 diabetes mellitus
* Patients must have bilateral sensorimotor distal peripheral neuropathy attributable to diabetes mellitus
* Patients must have blood glucose control measured as HbA1c=<11%
* Patients must be 18 years of age or older.
* Patients must be able to return to all follow-up visits

Exclusion Criteria:

* Patients must not have symptoms of diabetic peripheral neuropathy that cannot be distinguished from other etiologies
* Patients must not have a neurologic disease or neuropathy from a cause other than diabetes mellitus that would interfere with correct evaluation of symptomatic peripheral neuropathy.
* Patient currently has uncontrolled high blood pressure
* You have other medical problems that your doctor feels would make it unsafe for you to participate in this study such as liver or kidney problems
* You are a woman of childbearing age and unwilling or unable to use effective contraceptive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2004-10; Study Completion 2005-11

PRIMARY OUTCOMES:
The objectives of this study is to evaluate the effect of ruboxistaurin on subjects with diabetic peripheral polyneuropathy

SECONDARY OUTCOMES:
Ruboxistaurin will improve quantitative sensory testing and increase nerve fiber density in subjects with diabetic peripheral polyneuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Norfolk, Virginia, United States

REFERENCES:
- [Derived] Casellini CM, Barlow PM, Rice AL, Casey M, Simmons K, Pittenger G, Bastyr EJ 3rd, Wolka AM, Vinik AI. A 6-month, randomized, double-masked, placebo-controlled study evaluating the effects of the protein kinase C-beta inhibitor ruboxistaurin on skin microvascular blood flow and other measures of diabetic peripheral neuropathy. Diabetes Care. 2007 Apr;30(4):896-902. doi: 10.2337/dc06-1699. PMID 17392551